CLINICAL TRIAL: NCT00585780
Title: Prazosin to Reduce Stress-Induced Alcohol/Drug Craving and Relapse
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0705002691; 4R01AA020504-05 (NIH)
Record Dates: First submitted 2007-12-25; First posted 2008-01-03 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Prazosin

STUDY DESIGN:
Intervention Model Description: Interaction effects of Alcohol withdrawal distress with Prazosin versus Placebo effects during the trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization into Prazosin/Placebo treatment was conducted by the Yale Stress Center biostatistician using an Urn randomization procedure that balanced groups on gender, age, nicotine smoking status, education years and lifetime history of DSM-IVTR anxiety disorders, including Post Traumatic Stress Disorder (PTSD). Random assignment of each patient was provided to the Yale Investigational Drug Service (IDS) Pharmacist, who formulated identical, matched tablets of Prazosin and Placebo, and provided dosing in weekly blister packs labeled by day and time of dosing for each subject to study staff for dispensing. All study personnel, including investigators, physicians, study staff and patients remained blind to medication group.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Alcohol Withdrawal on Prazosin (Active Comparator): High AW was determined by those scoring at or above the median on Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) assessment. High AW were randomized to Prazosin 16 mg/day (tid) administered for 12 weeks with fish-bowl contingency management for weekly treatment attendance and manualized 12-Step relapse prevention counseling in a double blind manner.
  Interventions: Drug: Prazosin Tablet
- High Alcohol Withdrawal on PLA (Placebo Comparator): High AW was determined by those scoring at or above the median on Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) assessment. High AW were randomized to Placebo tablets administered tid for 12 weeks with fish-bowl contingency management for weekly treatment attendance and manualized 12-Step relapse prevention counseling in a double blind manner.
  Interventions: Drug: Placebo Tablet
- Low Alcohol Withdrawal on Prazosin (Active Comparator): Low AW was determined by those scoring below the median on Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) assessment. Low AW were randomized to Prazosin 16 mg/day (tid) administered for 12 weeks with fish-bowl contingency management for weekly treatment attendance and manualized 12-Step relapse prevention counseling in a double blind manner.
  Interventions: Drug: Prazosin Tablet
- Low Alcohol Withdrawal on PLA (Placebo Comparator): Low AW was determined by those scoring below the median on Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) assessment.Placebo tablets administered tid for 12 weeks with fish-bowl contingency management for weekly treatment attendance and manualized 12-Step relapse prevention counseling in a double blind manner.
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Prazosin Tablet — Target medication dosing was three times/day (t.i.d. dosing) with 5 mg in the morning, 5 mg in the afternoon and 6 mg at night reached at the end of the 2-week period, and maintained at this or their highest tolerated dose until week 11, followed by a 5-day taper in week 12, as in previous research.The titration schedule was as follows: 1 mg dose at bedtime for 2 nights, followed by a 1mg dose morning and night (8 AM/8 PM) on day 3, then 2 mg dose t.i.d., on days 4-6, 3 mg dose (2 pills each) morning and afternoon, and 4 mg dose (2 pills) at night for days 7-9, increased to 4 mg dosing t.i.d. on days 10-13, and from day 14 through week 11, 5 mg (1 pill) each in the morning and afternoon, and 6 mg for the night (2 pills) dose. This was followed by a 5-day taper in week 12. Patients were initiated on study medication upon presenting with a negative breathalyzer without any minimum pre-treatment alcohol abstinence period prior to medication initiation.
  Arms: High Alcohol Withdrawal on Prazosin; Low Alcohol Withdrawal on Prazosin
Drug: Placebo Tablet — Placebo tablets identical in appearance and dosing schedule as the active study medication was utilized
  Arms: High Alcohol Withdrawal on PLA; Low Alcohol Withdrawal on PLA

SUMMARY:
To test the preliminary efficacy of 16.0 mg of Prazosin daily versus placebo in treatment seeking alcohol dependent individuals. This proposal is a laboratory and treatment outcome study to examine the effects of Prazosin on brief exposure to stress, drug cues and neutral situations on alcohol and drug craving, mood and neurobiological reactivity in a sample of cocaine and/or alcohol dependent individuals. Prazosin will be beneficial for reduction in stress and alcohol cue induced craving and related arousal. In a sample of treatment-seeking alcohol dependent men and women, we propose to examine (a) differences in measures of alcohol craving, emotion state, hypothalamic-pituitary-adrenal (HPA) activation, physiological arousal and plasma catecholamine response to stress imagery and to alcohol cue imagery as compared to neutral imagery; (b) reduction in alcohol abstinence symptoms; and (c) improvement in alcohol treatment outcomes as measured by reductions in heavy drinking days, any drinking days, secondarily on drinks/day, anxiety, mood and sleep.

DETAILED DESCRIPTION:
This is a proof-of-concept (POC) experimental therapeutics study with 2 arms. The first is a double-blind placebo controlled laboratory study with 40 individuals meeting current alcohol dependence criteria (DSM-IVTR) who are admitted to the Clinical Neuroscience Research Unit and initiated on Prazosin vs Placebo (16mg/day) after admission and initial detoxification (if required). Experimental laboratory sessions are conducted after subjects achieved full dose after the 2-week titration, in week 3-4 of inpatient stay. The laboratory outcomes included alcohol craving, anxiety, negative affect and neuroendocrine and sympathetic arousal measures. Individuals who wished to remain on study medication for the outpatient (Arm 2) were maintained on study medication throughout the outpatient phase for a total period of 12 weeks.

Arm 2 of the POC study is a 12-week randomized clinical trial (RCT) of Prazosin (16mg/day) versus Placebo in 100 treatment seeking alcohol dependent individuals, to assess whether high anxiety and distress, including alcohol craving, manifest as increased alcohol withdrawal symptoms at treatment entry moderates Prazosin effects on alcohol use outcomes. Primary alcohol use outcomes include heavy drinking days, any drinking days and secondarily drinks/day. Additional secondary outcomes include alcohol craving, anxiety and mood symptoms and sleep disturbances. Patients from Arm 1 who wished to continue on study medication for the outpatient phase were included in Arm 2. Arm 2 patients were initiated on study medication upon presenting with a negative breathalyzer without any minimum pre-treatment alcohol abstinence period prior to medication initiation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals, ages 18-70 with alcohol dependence, treatment seeking with varying levels of alcohol withdrawal symptoms.
* meet current DSM-IV criteria for alcohol dependence,
* Subject has voluntarily given informed consent and signed the informed consent document.
* Able to read English and complete study evaluations.

Exclusion Criteria:

* Meet current criteria for dependence on another psychoactive substance, excluding nicotine and caffeine;
* Any current use of opiates;
* Current use of any psychoactive drugs, including anxiolytics, antidepressants, naltrexone or disulfram, except for stabilized on SSRIs
* Any psychotic disorder or current Axis I psychiatric symptoms requiring specific attention, including need for psychiatric medications for current major depression and anxiety disorders
* Significant underlying medical conditions such as cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude patient from fully cooperating or be of potential harm during the course of the study;
* Hypotensive individuals with sitting blood pressure below 90/60 mmHG.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2018-08 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine: Yale Stress Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Alcohol Withdrawal on Prazosin: High AW (Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) scores at or above 3 randomized to Prazosin 16 mg/day (tid) for 12 weeks.
- High Alcohol Withdrawal on PLA: High AW (Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) scores at or above 3 randomized to matching Placebo tablets (tid) for 12 weeks.
- Low Alcohol Withdrawal on Prazosin: Low AW (Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) scores at or below 3 randomized to Prazosin 16 mg/day (tid) for 12 weeks.
- Low Alcohol Withdrawal on PLA: Low AW (Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) scores at or below 2 randomized to matching Placebo tablets (tid) for 12 weeks.
Period: Overall Study
Arm/Group | High Alcohol Withdrawal on Prazosin | High Alcohol Withdrawal on PLA | Low Alcohol Withdrawal on Prazosin | Low Alcohol Withdrawal on PLA
Started | 21 | 23 | 34 | 22
Completed | 13 | 14 | 21 | 14
Not Completed | 8 | 9 | 13 | 8

BASELINE CHARACTERISTICS:
Population: Alcohol dependent individuals (men and women) between the ages of 18-70, evaluated using CIWA-Ar for alcohol withdrawal symptoms to be included in High and Low alcohol withdrawal categories.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Alcohol Withdrawal on Prazosin | High Alcohol Withdrawal on PLA | Low Alcohol Withdrawal on Prazosin | Low Alcohol Withdrawal on PLA | Total
Number analyzed (Participants) | 21 | 23 | 34 | 22 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (9.8) | 39.2 (11.1) | 39.6 (10.8) | 41.4 (11.9) | 40.65 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 13 | 7 | 35
  Male | 13 | 16 | 21 | 15 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12 | 10 | 20 | 9 | 51
  African American | 9 | 13 | 14 | 12 | 48
  Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heavy Drinking Days (HDD%) During the Full Dose Period From Weeks 3-12
Description: Percentage of heavy drinking days (HDD%) during the full dose period from weeks 3-12 where heavy drinking day (HDD) is defined as 5 or more for men and 4 or more for women in one sitting, measured as yes (1) or no(0), assessed via self reports by daily surveys and time-line follow back assessments
Time Frame: daily over 12 weeks
Population: Mean percentage of heavy drinking days (HDD%) during the full dose period from weeks 3-12
Measure: Mean (Standard Error); unit: percentage of heavy drinking days
Groups:
- High Alcohol Withdrawal (AW) on Prazosin: High AW (Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) scores at or above 3 randomized to Prazosin 16 mg/day (tid) for 12 weeks.
- High Alcohol Withdrawal (AW) on PLA: High AW (Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) scores at or above 3 randomized to matching Placebo tablets (tid) for 12 weeks.
- Low Alcohol Withdrawal (AW) on Prazosin: Low AW (Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) scores at or below 3 randomized to Prazosin 16 mg/day (tid) for 12 weeks.
- Low Alcohol Withdrawal (AW) on PLA: Low AW (Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) scores at or below 2 randomized to matching Placebo tablets (tid) for 12 weeks.
Arm/Group | High Alcohol Withdrawal (AW) on Prazosin | High Alcohol Withdrawal (AW) on PLA | Low Alcohol Withdrawal (AW) on Prazosin | Low Alcohol Withdrawal (AW) on PLA
Number analyzed (Participants) | 21 | 23 | 34 | 22
percentage of heavy drinking days | 8.2 (4.09) | 27.11 (7.97) | 31.29 (7.42) | 7.32 (3.54)
Statistical Analysis 1: Comparison: High Alcohol Withdrawal (AW) on Prazosin vs High Alcohol Withdrawal (AW) on PLA; Intent-to-treat (ITT) analyses with baseline AW severity (mean-centered continuous CIWA-Ar scores) as a moderator of Time (Pre-Full Dose(FD): weeks 1-2; Post FD: weeks 3-12) were conducted with linear or generalized linear mixed effect (LME/GLME) piecewise growth models for continuous and binary outcomes. Control variables that were modeled in all analyses. As hypothesized, significant interactions were tested using AW median cut-offs for high and Low AW groups; Test type: Other — Expected outcome was that Prazosin will be better than placebo in reducing HDD% among High AW individuals but no differences by medication treatment in the Low AW individuals; p = 0.016, Mixed Models Analysis — This is for the apriori hypothesis of significant AWX Treatment X Time effect; Simple effects were conducted to assess source of the interaction; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.1 to 0.55]

2. Primary Outcome: Percent of Drinkings Days During the Full Dose Period Between Weeks 3 and 12
Description: Percent of any drinkings days over the full dose period from weeks 3 to 12, defined as any alcoholic drink consumed each day measured as yes (1) or no(0), assessed via self reports by daily surveys and time-line follow back assessments
Time Frame: daily over 12 weeks
Measure: Mean (Standard Error); unit: Mean percent of any drinking days
Arm/Group | High Alcohol Withdrawal on Prazosin | High Alcohol Withdrawal on PLA | Low Alcohol Withdrawal on Prazosin | Low Alcohol Withdrawal on PLA
Number analyzed (Participants) | 21 | 23 | 34 | 22
Mean percent of any drinking days | 26.89 (7.45) | 41.21 (9.36) | 53.35 (7.74) | 23.71 (6.90)
Statistical Analysis 1: Comparison: High Alcohol Withdrawal on Prazosin vs High Alcohol Withdrawal on PLA; [analysis description as in outcome 1, analysis 1]; Test type: Other — Expected outcome was that Prazosin will be better than placebo in reducing percent of drinking days (DD%) among High AW individuals but no differences by medication treatment in the Low AW individuals; p = 0.002, Mixed Models Analysis — This is for apriori hypothesized significant AW X Treatment X Post-full dose time interaction effect; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.28 to 0.92]

ADVERSE EVENTS:
Time Frame: Adverse event data obtained weekly for 12 week treatment period using a modified version of the Systematic Assessment for Treatment Emergent Effects (SAFTEE) assessing expected and unexpected side effects and serious adverse events.
Groups:
- High Alcohol Withdrawal on Prazosin: High AW scoring at or above 3 on Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) assessment randomized to Prazosin 16 mg/day (tid) administered for 12 weeks.
  Prazosin Tablet: Target medication dosing was three times/day (t.i.d. dosing) with 5 mg in the morning, 5 mg in the afternoon and 6 mg at night reached at the end of the 2-week period, and maintained at this or their highest tolerated dose until week 11, followed by a 5-day taper in week 12, as in previous research.
- High Alcohol Withdrawal on PLA: High AW scoring at or above 3 on Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) assessment randomized to Placebo tablets administered tid for 12 weeks in a double blind manner.
  Placebo Tablet: Placebo tablets identical in appearance and dosing schedule as the active study medication was utilized
- Low Alcohol Withdrawal on Prazosin: Low AW scoring at or below 2 on Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) assessment randomized to Prazosin 16 mg/day (tid) administered for 12 weeks in a double blind manner.
  Prazosin Tablet: Target medication dosing was three times/day (t.i.d. dosing) with 5 mg in the morning, 5 mg in the afternoon and 6 mg at night reached at the end of the 2-week period, and maintained at this or their highest tolerated dose until week 11, followed by a 5-day taper in week 12, as in previous research.
- Low Alcohol Withdrawal on PLA: Low AW scoring at or below 2 on Clinical Institute of Withdrawal for Alcohol Revised (CIWA-Ar) assessment and randomized to Placebo tablets administered tid for 12 weeks in a double blind manner.
  Placebo Tablet: Placebo tablets identical in appearance and dosing schedule as the active study medication was utilized
Arm/Group | High Alcohol Withdrawal on Prazosin | High Alcohol Withdrawal on PLA | Low Alcohol Withdrawal on Prazosin | Low Alcohol Withdrawal on PLA
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23 | 0/34 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23 | 1/34 | 1/22
Other Adverse Events (participants affected / at risk) | 4/21 | 3/23 | 9/34 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Alcohol Withdrawal on Prazosin (N=21) | High Alcohol Withdrawal on PLA (N=23) | Low Alcohol Withdrawal on Prazosin (N=34) | Low Alcohol Withdrawal on PLA (N=22)
Alcohol intoxication (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 — Patient was admitted overnight after arriving at the ER with a blood alcohol concentration of 49mg/dl. Patient was referred back to the clinic the next morning to engage in treatment.
weakness and fainting (Social circumstances) | 0 | 0 | 0 | 1 (1) — Patient was admitted to the ER overnight after complaints of feeling faint and weakness with reports of being stressed and overwhelmed.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Alcohol Withdrawal on Prazosin (N=21) | High Alcohol Withdrawal on PLA (N=23) | Low Alcohol Withdrawal on Prazosin (N=34) | Low Alcohol Withdrawal on PLA (N=22)
Ligtheadedness/dizzy (Cardiac disorders) | 1 (2) | 1 (1) | 2 (4) | 1 (1) — Dizzy and/or lightheadedness
Pain (Nervous system disorders) | 2 (6) | 1 (3) | 4 (4) | 2 (7) — subjective rating of pain
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 2 (4) | 2 (4) — subjective reporting of headache
Cold and Flu (Infections and infestations) | 1 (5) | 2 (4) | 3 (4) | 2 (2) — Patient report of cold and flu-like symptoms

LIMITATIONS AND CAVEATS:
There was not adequate power to assess sex differences, and specific sensitivity and specificity data for apriori AW cutoffs for Prazosin benefit in high AW group needs to be determined in future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT00585780/Prot_SAP_000.pdf